CLINICAL TRIAL: NCT04584619
Title: Clariance Idys™ TLIF 3DTi Device Prospective Post Market Clinical Follow-up
Brief Title: Idys™ TLIF 3DTi Post Market Clinical Follow-up
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Clariance (Industry)
Responsible Party: Sponsor
Other Study IDs: 31PMCF-DrG
Record Dates: First submitted 2020-09-30; First posted 2020-10-14 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Degenerative Disc Disease; Grade 1 Spondylolisthesis
Keywords: Spine; Interbody fusion device
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Spine fusion surgery with Clariance Idys TLIF 3DTi — Posterior fusion of the lumbar spine with Clariance Idys TLIF 3DTi interbody fusion device used in conjunction with a posterior fixation system (pedicle screws and rod).

SUMMARY:
The aim of this observational post-marketing study is to provide additional information on the safety and effectiveness of Idys™ TLIF 3DTi at up to 24 months post transforaminal lumbar fusion in usual surgical practice.

DETAILED DESCRIPTION:
The primary endpoint is to evaluate the effectiveness of the Idys™ TLIF (Transforaminal Lumbar Interbody Fusion) 3DTi (Porous Titanium additive manufacturing) by measuring the evolution of the rate of fusion during the postoperative period.

The secondary endpoints are to analyze the safety and the patient's benefit of the Idys™ TLIF 3DTi by evaluating several point of view:

* The adverse events related to the surgery;
* The functional improvement between preoperative state and the different follow-up time points using the Oswestry Disability Index (ODI);
* The improvement of back pain between preoperative state and the different follow-up time points using the Visual Analog Scale (VAS) (legs and back);
* The evolution of several radiologic lumbar parameters to assess the correction and its stability.

ELIGIBILITY:
Inclusion Criteria:

* English Speaking patients
* Patient with skeletal maturity
* Patient with

  * degenerative disc disease at one or two levels from L2 to S1 and/or
  * grade 1 spondylolisthesis
* Surgical treatment with Idys TLIF 3DTi interbody fusion device used in conjunction with a posterior fixation system (pedicle screws and rod).

Exclusion Criteria:

* Off-label indications.
* Any medical or surgical condition which would preclude the potential benefit of spinal implant surgery.
* Any patient having a prior fusion at the level to be treated.
* Any patient being vulnerable
* Non-English speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who need fusion of spinal lumbar segments
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Evolution of the Fusion rate | 6 months, 12 months, 24 months postoperatively
  Evolution of the radiological assessment of bony fusion at 3 different time point

SECONDARY OUTCOMES:
Adverse events | Up to 24 months postoperatively
  To quantify and describe adverse events
Evolution of the Patient Disability | Preoperatively and then 6 weeks, 6 months, 12 months and 24 months postoperatively
  Assessment, at different time points, of the disability using Oswestry Disability Index score (range 0 to 100 with zero corresponding to no disability and 100 corresponding to the maximum disability possible)
Evolution of the Patient Pain | Preoperatively and then 6 weeks, 6 months, 12 months and 24 months postoperatively
  Assessment, at different time points, of the pain using Visual Analogue Scale (range 0 to 10 with higher scores meaning a worse outcome)
Radiologic Outcomes - Evolution of the lordosis angles (degree) | Preoperatively and then 6 weeks, 6 months, 12 months and 24 months postoperatively
  Measurements, on x-rays at different time points, of the lordosis angle at pathological / implanted level and of the global lordosis angle between L1/S1
Radiologic Outcomes - Evolution of the Intervertebral Height (mm) | Preoperatively and then 6 weeks, 6 months, 12 months and 24 months postoperatively
  Measurements, on x-rays at different time points, of the anterior and the posterior inter-vertebral height.
Radiologic Outcomes - Stability of the Idys TLIF 3DTi Device | 6 weeks, 6 months, 12 months and 24 months postoperatively
  Measurement ,on x-rays at different time points, of the anterior position of the Idys TLIF 3DTi device

CONTACTS AND LOCATIONS:
Overall Officials: Mukund Gundanna, Dr, Principal Investigator — Brazos Spine
Locations (1):
- Brazos Spine, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No